CLINICAL TRIAL: NCT01001819
Title: DNA Microarray Analysis of Gene Expression in Chronic Rhinosinusitis
Status: Completed | Type: Observational
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Marvin Fried, Professor, Otorhinolaryngology, Montefiore Medical Center
Other Study IDs: 05-01-005E
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Chronic Rhinosinusitis w/o Nasal Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Chronic Rhinosinusitis w/o nasal polyps
- 2: No sinus disease

SUMMARY:
Analysis of differential gene expression in patients with chronic rhinosinusitis without polyps compared to unaffected patients. Correlation of abnormal gene expression with surgical outcomes.

ELIGIBILITY:
Affected patients:

* Two or more of the following symptoms should be present for 12 weeks or more: anterior mucopurulent drainage, posterior mucopurulent drainage; nasal obstruction; and facial pain-pressure-fullness.

  * Signs of nasal inflammation such as discolored mucus, edema of the middle meatus or ethmoid area should be documented by endoscopy.
  * The symptoms of rhinosinusitis have failed to resolve or have recurred after a treatment course with antibiotics and nasal and/or oral steroids.
  * The diagnosis of rhinosinusitis should be confirmed with a CT scan.
  * Patients deny recent (within one year) cigarette smoking or exposure to inhaled substances that are potentially harmful to respiratory epithelium
  * Patients were not previously diagnosed with reactive airway disease or aspirin sensitivity.
  * Patients also must meet the standard criteria for endoscopic sinus surgery and scheduled to undergo their procedure at MMC.

Unaffected Patients:

Patients undergoing elective nasal surgery at MMC.

* Patients deny symptoms of allergic rhinitis such as nasal congestion, nasal discharge, itching, sneezing.
* Patients deny symptoms of chronic or acute rhinosinusitis such as nasal obstruction, facial pain-fullness-pressure, anosmia, anterior and/or posterior mucopurulent drainage.
* Nasal endoscopy showed no evidence of nasal inflammatory disease, such as erythema, edema, polyps, or discolored mucus.
* Patients do not have history of prior sinus surgeries and were not previously diagnosed with CRS.

  1. Patients deny recent (within one year) cigarette smoking or exposure to inhaled substances that are potentially harmful to respiratory epithelium.
  2. Patients were not diagnosed with reactive airway disease or aspirin sensitivity.
* The absence of evidence of inflammation, such as inflammatory infiltrate or epithelial dysplasia on histopathologic exam of nasal mucosa obtained during surgical procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Chronic Rhinosinusitis w/o nasal polyps who meet eligibilty requirements and are undergoing sinus surgery and patients w/o sinus disease who are undergoing intranasal surgery and meet eligbility requirements
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2005-03; Primary Completion 2008-11-18 (Actual); Study Completion 2008-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marvin P Fried, MD, Principal Investigator — Montefiore Medical Center/Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States